CLINICAL TRIAL: NCT00834418
Title: A Relative Bioavailability Study of 20 mg Leflunomide Tablets Under Fasting Conditions
Brief Title: Leflunomide 20 mg Tablets Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: R02-561
Record Dates: First submitted 2009-01-30; First posted 2009-02-03 (Estimated); Results first posted 2009-08-18 (Estimated); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — Leflunomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Leflunomide (Experimental): Leflunomide 20 mg Tablet
  Interventions: Drug: Leflunomide 20 mg Tablets
- Arava™ (Active Comparator): Arava™ 20 mg Tablet
  Interventions: Drug: ARAVA™ 20 mg Tablets

INTERVENTIONS:
Drug: Leflunomide 20 mg Tablets — 1 x 20 mg, single-dose fasting
  Arms: Leflunomide
Drug: ARAVA™ 20 mg Tablets — 1 x 20 mg, single-dose fasting
  Arms: Arava™

SUMMARY:
This study will compare the relative bioavailability (rate and extent of absorption) of 20 mg Leflunomide Tablets by TEVA Pharmaceuticals Industries, Ltd. with that of 20 mg ARAVA™ Tablets by Aventis Pharmaceuticals, Inc. following a single oral dose (1 x 20 mg tablet) in healthy adult subjects under fasting conditions.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA bioequivalence statistical methods

ELIGIBILITY:
Inclusion Criteria:

* Screening Demographics: All subjects selected for this study will be healthy men or women 18 years of age or older at the time of dosing. The weight range will not exceed ± 20% for height and body frame as per Desirable Weights for Adults - 1983 Metropolitan Height and Weight Table.
* Screening procedures: Each subject will complete the screening process within 28 days prior to dosing. Consent documents for both the screening evaluation and HIV antibody determination will be reviewed, discussed, and signed by each potential participant before full implementation of screening procedures.
* Screening will include general observations, physical examination, demographics, medical and medication history, an electrocardiogram, sitting blood pressure and heart rate, respiratory rate and temperature. The physical examination will include, but may not be limited to, an evaluation of the cardiovascular, gastrointestinal, respiratory and central nervous systems.
* The screening clinical laboratory procedures will include:

  1. Hematology: hematocrit, hemoglobin, WBC count with differential, RBC count, platelet count;
  2. Clinical Chemistry: serum creatinine, BUN, glucose, AST(GOT), ALT(GPT), albumin, total bilirubin, total protein, and alkaline phosphatase;
  3. HIV antibody and hepatitis B surface screens;
  4. Urinalysis: by dipstick; full microscopic examination if dipstick positive; and
  5. Urine Drug Screen: ethyl alcohol, amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine metabolites, opiates and phencyclidine.
  6. Serum Pregnancy Screen (female subjects only)
  7. Follicle Stimulating Hormone [FSH] (females only to verify postmenopausal status)
* If male must be vasectomized (at least 3 months)
* If female and:

  1. is postmenopausal for at least 1 year; or
  2. is surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy).

Exclusion Criteria:

* Subjects with a recent history of drug or alcohol addiction or abuse.
* Subjects with the presence of a clinically significant disorder involving the cardiovascular, respiratory, renal, gastrointestinal, immunologic, hematologic, endocrine, or neurologic system(s) or psychiatric disease (as determined by the clinical investigators).
* Subjects whose clinical laboratory test values are outside the accepted reference range and when confirmed on re-examination are deemed to be clinically significant.
* Subjects demonstrating a positive hepatitis B surface antigen screen or reactive HIV antibody screen.
* Subjects demonstrating a positive drug abuse screen when screened for this study.
* Female subjects who are currently breastfeeding.
* Female subjects demonstrating a positive pregnancy screen.
* Subjects with a history of allergic response(s) to leflunomide or related drugs.
* Subjects with a history of clinically significant allergies including drug allergies.
* Subjects with a clinically significant illness during the 4 weeks prior to dosing (as determined by the clinical investigators).
* Subjects who have taken any drug known to induce or inhibit hepatic drug metabolism in the 30 days prior to dosing.
* Subjects who report donating greater than 150 mL of blood within 30 days prior to dosing. All subjects will be advised not to donate blood for four weeks after completing the study.
* Subjects who have donated plasma (e.g. plasmapheresis) within 14 days prior to dosing. All subjects will be advised not to donate plasma for four weeks after completing the study.
* Subjects who report receiving any investigational drug within 30 days prior to dosing.
* Subjects who report taking any prescription medication in the 14 days prior to dosing, with the exception of postmenopausal women on HRT may continue their HRT and topical products without systemic absorption.
* Subjects who report an intolerance of direct venipuncture.
* Subjects who report consuming an abnormal diet during the 28 days prior to dosing.
* Subjects who report taking any product containing leflunomide within 180 days of dosing.
* Subjects who report taking any herbal products within 7 days prior to dosing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2002-06; Primary Completion 2002-07 (Actual); Study Completion 2002-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James D. Carlson, Pharm.D., Principal Investigator — PRACS Institute, Inc.
Locations (1):
- PRACS Institute, Ltd., Fargo, North Dakota, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Leflunomide | Arava™
Started | 42 | 42
Completed | 42 | 40
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Leflunomide | Arava™ | Total
Number analyzed (Participants) | 42 | 42 | 84
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 38 | 38 | 76
  >=65 years | 4 | 4 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 34 | 66
  Male | 10 | 8 | 18
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 40 | 40 | 80
  Hispanic | 1 | 2 | 3
  American Indian | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 42 | 42 | 84

OUTCOME MEASURES:

1. Primary Outcome: Cmax - Maximum Observed Concentration - Metabolite A77 1726 in Plasma
Description: Bioequivalence based on Cmax
Time Frame: Blood samples collected over 72 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Leflunomide | Arava™
Number analyzed (Participants) | 42 | 40
ng/mL | 2109.286 (407.044) | 1974.000 (421.291)
Statistical Analysis 1: Comparison: Leflunomide vs Arava™; Test type: Non-Inferiority or Equivalence — Analysis of variance (ANOVA) was performed on pharmacokinetic parameters of AUC0-72 and Cmax; Geometric Test/Ref Ratio x 100 = 107, 90% CI [99.6 to 116] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

2. Primary Outcome: AUC0-72 - Area Under the Concentration-time Curve From Time Zero to 72 Hours Post-dose - Metabolite A77 1726
Description: Bioequivalence based on AUC0-72
Time Frame: Blood samples collected over 72 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Leflunomide | Arava™
Number analyzed (Participants) | 42 | 40
ng*h/mL | 105806.888 (19068.308) | 103905.901 (19933.702)
Statistical Analysis 1: Comparison: Leflunomide vs Arava™; Test type: Non-Inferiority or Equivalence — Analysis of variance (ANOVA) was performed on pharmacokinetic parameters of AUC0-72 and Cmax; Geometric Test/Ref Ratio x 100 = 102, 90% CI [95.2 to 109] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigator is not permitted to discuss or publish trial results.